CLINICAL TRIAL: NCT00492063
Title: A Phase III, Observer-Blind, Randomized, Multi-Center Study to Evaluate Safety, Tolerability and Immunogenicity of a Single Intramuscular Dose of a Trivalent Subunit Influenza Vaccine Produced in Mammalian Cell Culture and of a Trivalent Subunit Influenza Vaccine Produced in Embryonated Hen Eggs, in Healthy Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Cell Culture-derived Influenza Vaccine in Healthy Adults and Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58P4
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Influenza
Keywords: safety; immunogenicity; non-inferiority; MDCK; cell culture-derived; subunit influenza vaccine; influenza prevention
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cell culture-derived influenza vaccine (cTIV) (Experimental)
  Interventions: Biological: Cell culture-derived trivalent subunit influenza vaccine (cTIV)
- Egg-derived influenza virus vaccine (TIV) (Active Comparator)
  Interventions: Biological: Egg-derived trivalent subunit influenza vaccine (TIV)

INTERVENTIONS:
Biological: Cell culture-derived trivalent subunit influenza vaccine (cTIV) — One vaccination (0.5 mL) of cell culture-derived influenza vaccine (cTIV) was administered in the deltoid muscle
  Arms: Cell culture-derived influenza vaccine (cTIV)
Biological: Egg-derived trivalent subunit influenza vaccine (TIV) — One vaccination (0.5 mL) of egg-derived influenza virus vaccine (TIV) was administered in the deltoid muscle
  Arms: Egg-derived influenza virus vaccine (TIV)

SUMMARY:
The present study aims to evaluate the safety and immunogenicity of the new influenza subunit vaccine produced in Madin Darby Canine Kidney (MDCK) cells in healthy adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years of age (first age group) OR over 60 years of age (second age group)
2. mentally competent to understand the nature, the scope and the consequences of the study
3. able and willing to give written informed consent prior to study entry
4. available for all the visits scheduled in the study
5. residence in the study area
6. in good health as determined by:

   1. medical history,
   2. physical examination,
   3. clinical judgment of the investigator.

Exclusion Criteria:

1. unable or unwilling to give written informed consent to participate in the study
2. suffering from an acute infectious disease
3. any serious disease such as:

   1. cancer (except for benign or localized skin cancer and non metastatic prostate cancer not currently treated with chemotherapy),_
   2. autoimmune disease (including rheumatoid arthritis),
   3. advanced arteriosclerotic disease or complicated diabetes mellitus,
   4. chronic obstructive pulmonary disease (COPD) requiring oxygen therapy,
   5. acute or progressive hepatic disease,
   6. acute or progressive renal disease,
   7. congestive heart failure
4. surgery planned during the study period
5. bleeding diathesis
6. history of hypersensitivity to any component of the study medication or chemically related substances, such as allergy to eggs or egg products
7. known or suspected impairment/alteration of immune function resulting from:

   1. receipt of immunosuppressive therapy (any cortical steroid or cancer chemotherapy),
   2. receipt of immunostimulants,
   3. receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study,
   4. high risk for developing an immunocompromising disease within the past 6 months
8. history of drug or alcohol abuse
9. laboratory confirmed influenza disease in the past 6 months
10. received influenza vaccine within the past 6 months
11. received another vaccine or any investigational agent within the past 60 days, or planned vaccination within 3 weeks following the study vaccination
12. any acute respiratory disease or infections requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis was acceptable) or experienced fever ≥ 38°C within the past 3 days
13. pregnant women or women who refused to use a reliable contraceptive method throughout the study (180 days)
14. any condition which, in the opinion of the investigator, might have interfered with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2654 (Actual)
Dates: Start 2004-09; Primary Completion 2004-12 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (5):
- Poland (5):
  - Wojewódzki Szpital Dzieciecy, Ul. Langiewicza 2, Kielce
  - N ZOZ Jagiellonskie, Centrum Medyczne Sp. z o.o., Os. Jagiellonskie 1, Kraków
  - Praktyka Grupowa Lekarzy POZ "Familia", Pl. Sikorskiego 6a, Kraków
  - Szpital Jana Pawła II, Ul. Pradnicka 80, Kraków
  - Centrum Farmakologii Klinicznej, Krakow

REFERENCES:
- [Result] Szymczakiewicz-Multanowska A, Groth N, Bugarini R, Lattanzi M, Casula D, Hilbert A, Tsai T, Podda A. Safety and immunogenicity of a novel influenza subunit vaccine produced in mammalian cell culture. J Infect Dis. 2009 Sep 15;200(6):841-8. doi: 10.1086/605505. PMID 19673651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 5 sites in Poland.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- cTIV (Adults): Subjects ≥18 to ≤60 years of age who received one vaccination of cell culture-derived influenza virus vaccine (cTIV)
- TIV (Adults): Subjects ≥18 to ≤60 years of age who received one vaccination of egg-derived influenza virus vaccine (TIV)
- cTIV (Elderly): Subjects ≥61 years of age who received one vaccination of cell culture-derived influenza virus vaccine (cTIV)
- TIV (Elderly): Subjects ≥61 years of age who received one vaccination of egg-derived influenza virus vaccine (TIV)
Period: Overall Study
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly)
Started | 652 | 648 | 678 | 676
Completed | 642 | 634 | 667 | 666
Not Completed | 10 | 14 | 11 | 10
Not completed — Death | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 5 | 4
Not completed — Lost to Follow-up | 6 | 11 | 5 | 3
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly) | Total
Number analyzed (Participants) | 652 | 648 | 678 | 676 | 2654
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (12.7) | 38.3 (13.3) | 69.1 (5.7) | 68.8 (5.6) | 54.0 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 376 | 371 | 389 | 375 | 1511
  Male | 276 | 277 | 289 | 301 | 1143

OUTCOME MEASURES:

1. Primary Outcome: Percentages Of Subjects Who Achieved HI Titer ≥40 After One Vaccination of Cell Culture-derived (cTIV) or Egg-derived (TIV) Influenza Subunit Vaccines
Description: Immunogenicity was measured as the percentage of adults (≥18 to ≤60 years) and elderly (≥61 years) achieving HI titers ≥40 at baseline (day 1) and three weeks (day 22) after one vaccination of cTIV or TIV vaccine for each of three vaccine strains, evaluated using the hemagglutination inhibition (HI) egg-derived antigen assay.
  In compliance with the requirements of the EMEA recommendations (CPMP/BWP/2490/00, CPMP/BWP/214/96), this criterion is met if the percentage of subjects achieving HI titers ≥40 is >70% in the ≥18 to ≤60 years of age group or >60% in the ≥61 years of age group.
Time Frame: Before vaccination (day 1) and three weeks after vaccination (day 22)
Population: Analysis was done on the per-protocol (PP) set, i.e. the subjects who received the vaccination correctly; provided evaluable data before and after vaccination; and with no major protocol violations, as defined before unblinding.
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly)
Number analyzed (Participants) | 650 | 644 | 672 | 674
Percentages
  A/H1N1 (Day 1) | 29 [26 to 33] | 33 [29 to 36] | 30 [27 to 34] | 31 [27 to 34]
  A/H1N1 (Day 22) | 92 [89 to 94] | 92 [89 to 94] | 85 [82 to 87] | 85 [82 to 88]
  A/H3N2 (Day 1) | 65 [61 to 69] | 63 [60 to 67] | 66 [63 to 70] | 59 [56 to 63]
  A/H3N2 (Day 22) | 99 [98 to 100] | 99 [98 to 99] | 97 [96 to 98] | 98 [97 to 99]
  B (Day 1) | 16 [13 to 19] | 18 [15 to 22] | 23 [20 to 26] | 20 [17 to 23]
  B (Day 22) | 90 [88 to 93] | 91 [88 to 93] | 90 [88 to 92] | 89 [87 to 91]
Statistical Analysis 1: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (HI titer ≥40) of cTIV to that of TIV vaccine for strain A/H1N1 after one vaccination in adults; Test type: Non-Inferiority or Equivalence — The percentage of subjects with HI titer ≥40 in the cTIV group is >10% lower than in the TIV group (i.e., the percentage of subjects with HI titer ≥40 in the cTIV group is non-inferior to that of TIV group if, for strain A/H1N1, the lower limit of the 95% CI of the difference in the percentages is greater than -10%); Group difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 2: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (HI titer ≥40) of cTIV to that of TIV vaccine for strain A/H3N2 after one vaccination in adults; Test type: Non-Inferiority or Equivalence — The percentage of subjects with HI titer ≥40 in the cTIV group is >10% lower than in the TIV group (i.e., the percentage of subjects with HI titer ≥40 in the cTIV group is non-inferior to that of TIV group if, for strain A/H3N2, the lower limit of the 95% CI of the difference in the percentages is greater than -10%); Group difference = 0, 95% CI 2-sided [-1 to 2]
Statistical Analysis 3: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (HI titer ≥40) of cTIV to that of TIV vaccine for strain B after one vaccination in adults; Test type: Non-Inferiority or Equivalence — The percentage of subjects with HI titer ≥40 in the cTIV group is >10% lower than in the TIV group (i.e., the percentage of subjects with HI titer ≥40 in the cTIV group is non-inferior to that of TIV group if, for strain B, the lower limit of the 95% CI of the difference in the percentages is greater than -10%); Group difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 4: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (HI titer ≥40) of cTIV to that of TIV vaccine for strain A/H1N1 after one vaccination in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Group difference = -1, 95% CI 2-sided [-4 to 3]
Statistical Analysis 5: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (HI titer ≥40) of cTIV to that of TIV vaccine for strain A/H3N2 after one vaccination in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Group difference = -1, 95% CI 2-sided [-2 to 1]
Statistical Analysis 6: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (HI titer ≥40) of cTIV to that of TIV vaccine for strain B after one vaccination in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; Group difference = 1, 95% CI 2-sided [-2 to 4]

2. Primary Outcome: Percentages Of Subjects Who Achieved Seroconversion Or Significant Increase In HI Titer After One Vaccination of cTIV or TIV
Description: Seroconversion or significant in HI titer is defined as the percentage of subjects with a prevaccination HI titer <10 (negative) to a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, at least a 4-fold increase in postvaccination HI titer. In compliance with the requirements of the EMEA recommendations (CPMP/BWP/2490/00, CPMP/BWP/214/96), the criterion is met if the percentage of subjects achieving seroconversion/significant increase is >40% in the ≥18 to ≤60 years of age group or >30% in the ≥61 years of age group.
Time Frame: Three weeks after vaccination (day 22)
Population: Analysis was performed on the PP set.
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly)
Number analyzed (Participants) | 650 | 644 | 672 | 674
Percentages
  A/H1N1 | 69 [65 to 73] | 67 [63 to 71] | 55 [51 to 59] | 55 [51 to 59]
  A/H3N2 | 63 [59 to 67] | 64 [60 to 68] | 68 [65 to 72] | 65 [61 to 69]
  B | 85 [82 to 87] | 81 [78 to 84] | 80 [77 to 83] | 73 [70 to 77]
Statistical Analysis 1: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (seroconversion or significant increase in HI titer) after one vaccination of cTIV to that of TIV vaccine for strain A/H1N1 in adults; Test type: Non-Inferiority or Equivalence — The percentage of subjects with seroconversion or significant increase in HI titer in the cTIV group is >10% lower than in the TIV group (i.e., the percentage of subjects with seroconversion or significant in HI titer of cTIV group is non-inferior to that of the TIV group if, for strain A/H1N1, the lower limit of the 95% CI of the difference in the percentages is greater than -10%); Group difference = 2, 95% CI 2-sided [-3 to 7]
Statistical Analysis 2: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (seroconversion or significant increase in HI titer) after one vaccination of cTIV to that of TIV vaccine for strain A/H3N2 in adults; Test type: Non-Inferiority or Equivalence — The percentage of subjects with seroconversion or significant increase in HI titer in the cTIV group is >10% lower than in the TIV group (i.e., the percentage of subjects with seroconversion or significant in HI titer of cTIV group is non-inferior to that of the TIV group if, for strain A/H3N2, the lower limit of the 95% CI of the difference in the percentages is greater than -10%); Group difference = -1, 95% CI 2-sided [-6 to 4]
Statistical Analysis 3: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (seroconversion or significant increase in HI titer) after one vaccination of cTIV to that of TIV vaccine for strain B in adults; Test type: Non-Inferiority or Equivalence — The percentage of subjects with seroconversion or significant increase in HI titer in the cTIV group is >10% lower than in the TIV group (i.e., the percentage of subjects with seroconversion or significant in HI titer of cTIV group is non-inferior to that of the TIV group if, for strain B, the lower limit of the 95% CI of the difference in the percentages is greater than -10%); Group difference = 4, 95% CI 2-sided [0 to 8]
Statistical Analysis 4: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (seroconversion or significant increase in HI titer) after one vaccination of cTIV to that of TIV vaccine for strain A/H1N1 in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Group difference = 0, 95% CI 2-sided [-6 to 5]
Statistical Analysis 5: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (seroconversion or significant increase in HI titer) after one vaccination of cTIV to that of TIV vaccine for strain A/H3N2 in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 2]; Group difference = 3, 95% CI 2-sided [-2 to 8]
Statistical Analysis 6: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (seroconversion or significant increase in HI titer) after one vaccination of cTIV to that of TIV vaccine for strain B in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 3]; Group difference = 6, 95% CI 2-sided [2 to 11]

3. Primary Outcome: Geometric Mean Ratio of Subjects After One Vaccination of cTIV or TIV
Description: Immunogenicity was measured as the geometric mean ratio (GMR), calculated as the ratio of postvaccination to prevaccination HI Geometric Mean Titers (GMTs), three weeks after (day 22) one vaccination of cTIV or TIV. In compliance with the requirements of the EMEA recommendations (CPMP/BWP/2490/00, CPMP/BWP/214/96), this criterion is met if the GMR (day 22/day 1) in HI antibody titer is >2.5 in the ≥18 to ≤60 years of age group or >2.0 in the ≥61 years of age group.
Time Frame: Three weeks after vaccination (day 22)
Population: Analysis was performed on the PP set.
Measure: Number (95% Confidence Interval); unit: Ratio
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly)
Number analyzed (Participants) | 650 | 644 | 672 | 674
Ratio
  A/H1N1 | 11 [10 to 13] | 11 [9.34 to 12] | 5.74 [5.15 to 6.41] | 5.96 [5.35 to 6.65]
  A/H3N2 | 5.99 [5.37 to 6.68] | 7.08 [6.34 to 7.9] | 7.25 [6.47 to 8.12] | 8.36 [7.46 to 9.36]
  B | 13 [12 to 15] | 12 [11 to 13] | 12 [11 to 13] | 9.29 [8.42 to 10]
Statistical Analysis 1: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (GMR) after one vaccination of cTIV to that of TIV vaccine for strain A/H1N1 in adults; Test type: Non-Inferiority or Equivalence — The value of GMR ratio of cTIV to TIV is >0.5 (i.e., the GMR of the cTIV group is non-inferior to that of the TIV group if, for strain A/H1N1, the lower limit of the 95% CI for ratio of GMRs at day 22 is greater than 0.5); Ratio of GMRs = 1.07, 95% CI 2-sided [0.9 to 1.28]
Statistical Analysis 2: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (GMR) after one vaccination of cTIV to that of TIV vaccine for strain A/H3N2 in adults; Test type: Non-Inferiority or Equivalence — The value of GMR ratio of cTIV to TIV is >0.5 (i.e., the GMR of the cTIV group is non-inferior to that of the TIV group if, for strain A/H3N2, the lower limit of the 95% CI for ratio of GMRs at day 22 is greater than 0.5); Ratio of GMRs = 0.85, 95% CI 2-sided [0.72 to 0.99]
Statistical Analysis 3: Comparison: cTIV (Adults) vs TIV (Adults); Non-inferiority testing in immune response (GMR) after one vaccination of cTIV to that of TIV vaccine for strain B in adults; Test type: Non-Inferiority or Equivalence — The value of GMR ratio of cTIV to TIV is >0.5 (i.e., the GMR of the cTIV group is non-inferior to that of the TIV group if, for strain B, the lower limit of the 95% CI for ratio of GMRs at day 22 is greater than 0.5); Ratio of GMRs = 1.14, 95% CI 2-sided [0.99 to 1.3]
Statistical Analysis 4: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (GMR) after one vaccination of cTIV to that of TIV vaccine for strain A/H1N1 in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of GMRs = 0.96, 95% CI 2-sided [0.82 to 1.12]
Statistical Analysis 5: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (GMR) after one vaccination of cTIV to that of TIV vaccine for strain A/H3N2 in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 2]; Ratio of GMRs = 0.87, 95% CI 2-sided [0.74 to 1.02]
Statistical Analysis 6: Comparison: cTIV (Elderly) vs TIV (Elderly); Non-inferiority testing in immune response (GMR) after one vaccination of cTIV to that of TIV vaccine for strain B in the elderly population; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 3]; Ratio of GMRs = 1.27, 95% CI 2-sided [1.11 to 1.4]

4. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions up to 7 Days After Vaccination
Description: The solicited local and systemic reactions were collected from day 1 up to and including day 7 after vaccination for both the vaccine groups.
Time Frame: Up to 7 days postvaccination
Population: Analysis was done on Safety population i.e., all subjects with vaccination and with some post-baseline safety data.
Measure: Number; unit: Number of Subjects
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly)
Number analyzed (Participants) | 652 | 648 | 678 | 676
Number of Subjects
  Ecchymosis | 18 | 22 | 26 | 25
  Erythema | 92 | 106 | 72 | 72
  Induration | 38 | 42 | 37 | 29
  Swelling | 25 | 27 | 23 | 17
  Pain | 141 | 111 | 64 | 32
  Chills | 25 | 29 | 23 | 26
  Malaise | 74 | 74 | 70 | 75
  Myalgia | 45 | 49 | 46 | 57
  Arthralgia | 31 | 27 | 41 | 44
  Headache | 81 | 79 | 69 | 70
  Sweating | 28 | 27 | 44 | 48
  Fatigue | 73 | 73 | 73 | 84
  Fever (≥38°C) | 2 | 5 | 5 | 5
  Stayed home due to reaction | 14 | 16 | 19 | 14
  Analgesic/antipyretic medication used | 44 | 40 | 34 | 29

ADVERSE EVENTS:
Time Frame: Throughout the study (day 1 to day 180)
Description: All serious adverse events (AEs) were collected throughout the study (day 1 to day 180).
Arm/Group | cTIV (Adults) | TIV (Adults) | cTIV (Elderly) | TIV (Elderly)
Serious Adverse Events (participants affected / at risk) | 7/652 | 5/648 | 19/678 | 18/676
Other Adverse Events (participants affected / at risk) | 261/652 | 257/648 | 224/678 | 207/676
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cTIV (Adults) (N=652) | TIV (Adults) (N=648) | cTIV (Elderly) (N=678) | TIV (Elderly) (N=676)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope Vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atherosclerosis obliterans (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | cTIV (Adults) (N=652) | TIV (Adults) (N=648) | cTIV (Elderly) (N=678) | TIV (Elderly) (N=676)
Injection site erythema (General disorders) | 92 (92) | 106 (106) | 72 (72) | 72 (72)
Injection site induration (General disorders) | 38 (38) | 42 (42) | 37 (37) | 29 (29)
Injection site pain (General disorders) | 141 (141) | 111 (111) | 64 (64) | 32 (32)
Malaise (General disorders) | 76 (76) | 75 (75) | 74 (74) | 76 (76)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (37) | 36 (36) | 48 (48) | 48 (48)
Myalgia (Musculoskeletal and connective tissue disorders) | 46 (46) | 51 (51) | 47 (47) | 58 (58)
Fatigue (General disorders) | 73 (73) | 73 (73) | 74 (74) | 85 (85)
Headache (Nervous system disorders) | 87 (87) | 88 (88) | 75 (75) | 75 (75)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 45 (45) | 48 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.